CLINICAL TRIAL: NCT03898804
Title: An Early Feasibility Study to Assess the Effects of the "Reconnecting the Hand and Arm to the Brain (ReHAB)" System
Brief Title: An Early Feasibility Study of the ReHAB System
Acronym: ReHAB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jennifer Sweet, MD (Other)
Responsible Party: Sponsor-Investigator, Jennifer Sweet, MD, Physician, University Hospitals Cleveland Medical Center
Organization: University Hospitals Cleveland Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: STUDY20190226
Record Dates: First submitted 2018-11-15; First posted 2019-04-02 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Tetraplegia
MeSH Terms: conditions — Quadriplegia

STUDY DESIGN:
Intervention Model Description: The study is a prospective, non-randomized, open-label, exploratory safety/feasibility trial of up to 12 subjects. The Primary Endpoint will be evaluation over the first 13 months after implantation, after which the subjects will have the option of removal of the device or continued participation in a long-term study for an additional 5 years, for a total of up to 73 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- BCI and FES (Experimental): Surgical implantation of the device and testing for 13 months with an optional 5 year extension study.
  Interventions: Device: BCI and FES

INTERVENTIONS:
Device: BCI and FES — The intervention consists of surgical implantation of the device components, BCI and FES that will interface with computers that process and decode neural information, compute stimulation parameters, and control communication between the device components. The device will be tested during research sessions spanning a 13-month period.

SUMMARY:
The purpose of this research study is to examine the feasibility of a system that involves implanting small electrodes in the parts of the brain that control movement and sensation, and combining that with electrodes in the upper arm and shoulder to activate paralyzed muscles of the arm and hand. This system is intended for people with extensive paralysis in their arms. The small electrodes in the brain will be used to attempt to measure intended movements, and the muscles in the arm and hand will be stimulated to attempt to follow those intentions.

The study is a prospective, non-randomized, open-label, exploratory safety/feasibility trial of up to 12 subjects. The Primary Endpoint will be evaluation over the first 13 months after implantation, after which the subjects will have the option of removal of the device or continued participation in a long-term study.

DETAILED DESCRIPTION:
The overall purpose of this trial is to advance development of a novel technological approach to allow individuals with tetraplegia to interact with their environment using their own paralyzed limbs by combining recording of brain activity, brain stimulation to provide sensory feedback, and stimulation of the paralyzed extremities based on neural recordings.

Device Name:

Reconnecting the Hand and Arm to the Brain (ReHAB) System

Intended Use The proposed device is intended to allow greater functional independence for individuals who are paralyzed due to disease or injury. The purpose of this trial is to advance development of a novel technological approach to allow individuals with tetraplegia to interact with their environment using their own paralyzed limbs by combining recording of brain activity, brain stimulation to provide sensory feedback, and stimulation of the paralyzed extremities based on neural recordings.

The target population are individuals with high tetraplegia, defined as less than antigravity weakness of both upper extremities and both lower extremities as a result of an identified and static (stable for at least 3 months) injury or disease affecting upper motor neurons process that prevents motor neural activity from activating muscles below the neck to perform functional activities. Injuries and diseases that lead to this clinical condition include spinal cord injury, and stroke.

Objective(s):

The primary objective of this study is to evaluate the safety, tolerability, and potential efficacy of an approach combining multiple intracortical brain recording/stimulating microarrays with direct peripheral nerve and muscle stimulation for restoration of arm and hand movement in people with high tetraplegia.

Secondary objectives include validation of the combined platform described above as a clinical device to allow paralyzed individuals to have a more meaningful interaction with their environment as assessed by ability to perform brain-controlled reaching and grasping tasks that ultimately might allow for greater functional independence.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 22 and 65 years of age.
2. Tetraplegia due to a static identified disease process (spinal cord injury or stroke) that prevents functional activity of the upper extremity.
3. Onset of tetraplegia at least 12 months prior to enrollment, with stability of weakness for at least 3 months.
4. Must have sufficiently intact cortical motor structures and stable medical prognoses to be able to perform the BCI control tasks for at least one year. .
5. Ability to speak understandably or, if unable to speak understandably, a reliable means of yes/no communication.
6. Life expectancy greater than 13 months.
7. Chronic care environment within a three-hour drive of the study site or the ability to temporarily relocate to a residence within a three-hour drive of the study site.
8. Willingness to remain available (geographically stable) for at least 13 months after enrollment, including maintenance of the evaluation schedule, frequent visits to the Investigator's office, and visits of Sponsor personnel to the subject's chronic care environment.
9. Willingness to allow videotape recordings to be made of the surgical procedure (for training purposes) and portions of the Feasibility Evaluations.
10. A stable psychosocial support system.
11. Scalp devoid of any lesions or skin breakdown precluding surgery.
12. Ability to provide voluntarily informed consent in accordance with Site institutional policies and willingness to release of Personal Health Information from the date of the injury or disease onset through the completion of the clinical Study.
13. Availability of caregivers capable of providing the necessary daily care of the subject's skin and electrode externalization sites.

Exclusion Criteria:

1. Presence of an implanted stimulator such as a pacemaker, spinal cord stimulator, cochlear implant, deep brain stimulator, vagus nerve stimulator, or defibrillator. (Implanted intrathecal pumps for pain or spasticity, cough implants, or diaphragmatic pacers are not excluded.)
2. Any active infection(s) or unexplained fever.
3. Active cancer within the one year prior to enrollment (other than adequately treated basal or squamous cell skin cancer).
4. Uncontrolled insulin-dependent diabetes mellitus.
5. Hydrocephalus requiring diversion of cerebrospinal fluid.
6. Autonomic dysreflexia within three months prior to enrollment that required urgent evaluation and pharmacologic intervention prescribed by a physician.
7. Seizure within 3 months prior to enrollment.
8. Any medical condition expected to require routine MRI imaging or subjects with contraindication(s) to MRI.
9. History of osteomyelitis or skin disorder that causes excessive skin sloughing, lesions or breakdown of the scalp.
10. Chronic use of medications such as sedatives that may significantly retard motor coordination and cognitive ability.
11. Chronic use of anticoagulant medications. (Subjects receiving prophylactic anticoagulation solely for the prevention of deep venous thrombosis are not excluded, but must be able to have their prophylactic anticoagulation suspended temporarily for the surgical procedure and immediate post-operative period.)
12. Chronic use of steroids or immunosuppressant therapy.
13. Active treatment for another serious medical, neurological or psychiatric disease or disorder that could seriously affect the subject's ability to undergo surgical implantation of the electrodes or participate in the testing sessions.
14. Pregnant, lactating, or of childbearing age and not using adequate birth control.
15. Active consumption of more than 1 alcoholic beverage per day.
16. Suicide attempt within 12 months prior to enrollment.
17. History of myocardial infarction or unstable cardiac arrhythmia.
18. Enrollment in any other investigational study that may interfere with the time commitments required of this study.
19. Subjects who are immunocompromised.
20. Subjects who require ongoing diathermy or ultrasound treatments.
21. Subjects with severe upper extremity joint contractures or Ashworth spasticity scores of 4 that would limit functional movements.
22. Subjects who have contraindication(s) to CT.
23. Subjects who are ventilator dependent. Subjects who are sometimes ventilator-assisted (for example, while sleeping) are not excluded.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-04-09 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-related adverse events | 13 months
  Successful implantation of brain and extremity recording/stimulating electrodes for 1 year without explantation or device-related serious adverse events.

SECONDARY OUTCOMES:
Success rate of target acquisition of a cursor on a computer screen controlled by neural signals, using a standard center-out-center random target display. | 13 months
  The participant will control the position of a cursor on a monitor using the recorded neural signals and attempt to move the cursor to the target.
Change in number of tasks performed as measured by the ADL Abilities Test. | 13 months
  The participant will control the stimulated movement of their arm and hand using the recorded neural signals. The participant will demonstrate the ability to perform some of the activities of daily living (ADLs) that are part of the ADL Abilities Test.
Change in number of objects successfully grasped and moved during a timed session, as measured by the Grasp Release Test. | 13 months
  The participant will control the stimulated movement of their arm and hand using the recorded neural signals. The participant will demonstrate the ability to grasp and move a series of objects that are part of the Grasp Release Test.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Sweet, M.D., Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gardner J. Savings for states? Senate budget aims to reinstate Medicaid cost sharing. Mod Healthc. 1997 Jul 14;27(28):66. No abstract available. PMID 10168522
- [Derived] Jakes RS, Alexander BJ, Marcu V, Ajiboye AB, Tyler DJ. A methodological framework for the efficient characterization of peripheral nerve stimulation parameters. J Neural Eng. 2025 Oct 27;22(5):056041. doi: 10.1088/1741-2552/ae0d31. PMID 41022103
- [Derived] Jakes RS, Alexander BJ, Marcu VI, Ajiboye AB, Tyler DJ. A Methodological Framework for the Efficient Characterization of Peripheral Nerve Stimulation Parameters. medRxiv [Preprint]. 2025 May 23:2025.03.29.25324704. doi: 10.1101/2025.03.29.25324704. PMID 40661284
- See also: This website provides information about the ReHAB Study. — https://rehabstudy.org